CLINICAL TRIAL: NCT06550960
Title: Evaluation of a Soft Tissue Biopsy System for Trans-rectal and Trans-perineal Biopsy of the Prostate Using Standard of Care and Artificial Intelligence (AI) Analysis
Brief Title: Evaluation of SureCore Plus Biopsy System
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Uro-1 Medical (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 23-01
Record Dates: First submitted 2024-07-30; First posted 2024-08-13 (Actual); Last update posted 2024-08-13 (Actual); Status verified 2024-07

CONDITIONS: BPH

STUDY DESIGN:
Intervention Model Description: Two-arm study of study biopsy needle and standard of care biopsy needle
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- SureCore Plus biopsy needle (Experimental): Prostate biopsy of subject with BPH with a SureCore biopsy needle
  Interventions: Device: Evaluation of two biopsy systems
- Standard of Care biopsy needle (Active Comparator): Prostate biopsy of subject with BPH with a standard of care (SOC) biopsy needle
  Interventions: Device: Evaluation of two biopsy systems

INTERVENTIONS:
Device: Evaluation of two biopsy systems — Each subject will have prostate biopsy taken in 6 locations in one lobe of the prostate and then biopsy in 6 locations in the other lobe of the prostate

SUMMARY:
This is a post-market study of a cleared biopsy system. The quality of tissue cores varies with standard of care biopsy needles. The SureCore Plus biopsy system is being evaluated as to quality and volume of tissue from prostate biopsy as compared to standard of care biopsy needles.

DETAILED DESCRIPTION:
Biopsy sampling of the prostate using TRUS or TPPB guidance is the current SoC approach for diagnosis of prostate cancer (CaP). Over the past decades the number of samples required and considered adequate has risen from 6 to 12-18 and sometimes as many as 30. Many practices routinely sample up to 20 cores of tissue. The SureCore Plus biopsy system is being to sample, obtain and retrieve prostate biopsy specimens in men undergoing scheduled diagnostic prostate biopsy and compare it with an standard of care (SoC) biopsy instrument and SoC method of specimen retrieval.

ELIGIBILITY:
Inclusion Criteria:

* Patient has BPH requiring a prostate biopsy
* Able and willing to provide consent

Exclusion Criteria:

* Active infection
* Subject participating in an other device study of the prostate

Ages: 18 Years to 80 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — This is biopsy of the prostate. Only males have a prostate.
Enrollment: 30 (Estimated)
Dates: Start 2024-08-05 (Estimated); Primary Completion 2024-12-31 (Estimated); Study Completion 2025-02-01 (Estimated)

PRIMARY OUTCOMES:
Procedure success | During the procedure
  > 3 mm/cc of tissue collected in each biopsy
Quality of biopsy tissue | During the procedure
  Ranking by pathologist on scale of 0=unable to read to 5=all tissue complete for reading. The higher scores mean a better outcome.

SECONDARY OUTCOMES:
Performance of the study device | During the procedure
  Ranking by MD using scale of 1=difficult to use to 5=outperformed SOC needles. The higher scores equate to better outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey Proctor, MD, Principal Investigator — Georgia Urology

IPD SHARING:
Plan to Share IPD: No